CLINICAL TRIAL: NCT01743651
Title: A Randomized, Double-Blind, Parallel Group Study to Compare the Safety and Efficacy Arbaclofen ER Tablets to Placebo and Baclofen Tablets, USP for the Treatment of Spasticity in Patients With Multiple Sclerosis
Brief Title: Efficacy Study of Arbaclofen to Treat Spasticity in Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Collaborators: Osmotica Pharmaceutical US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OS440-3002
Record Dates: First submitted 2012-11-28; First posted 2012-12-06 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2014-05

CONDITIONS: Spasticity; Multiple Sclerosis
Keywords: spasticity; multiple sclerosis; arbaclofen
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis | interventions — arbaclofen placarbil; Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Baclofen (Active Comparator): 80 mg/day of Baclofen Tablets, USP
  Interventions: Drug: baclofen
- Arbaclofen (Experimental): 40 mg/day of Arbaclofen Tablets
  Interventions: Drug: arbaclofen

INTERVENTIONS:
Drug: arbaclofen — 40 mg/day as 20 mg arbaclofen ER administered orally 2 times per day
  Other Names: OS440; AERT
  Arms: Arbaclofen
Drug: baclofen — 80 mg/day as 20 mg baclofen administered orally 4 times per day
  Arms: Baclofen
Drug: Placebo — arbaclofen image matched placebo tablets administered orally 2 times/day or baclofen image matched placebo capsules administered orally 4 times/day
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized (1:1:1), double-blind, active and placebo controlled, parallel group study to evaluate safety, tolerability and efficacy of oral arbaclofen in MS patients with spasticity.

Eligible subjects will be removed from anti-spasticity medications for at least one week and then begin study drug treatment with daily doses increasing up to the target dose which will then be maintained for at least 12 weeks. A down-titration will then occur over two weeks.

DETAILED DESCRIPTION:
This is a multicenter, randomized (1:1:1), double-blind, active and placebo controlled, parallel group study to evaluate safety, tolerability and efficacy of oral arbaclofen in MS patients with spasticity.

Eligible subjects will be removed from anti-spasticity medications for at least one week and then begin study drug treatment with daily doses increasing up to the target dose which will then be maintained for at least 12 weeks. A down-titration will then occur over two weeks with the final study visit occurring at 19 weeks from start of achieving the target dose or 22 weeks from the Study Visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) 18 to 65 years of age, inclusive, at the time of dosing
* Have an established diagnosis (per McDonald Criteria) of Multiple Sclerosis (either relapsing remitting or secondary progressive course), that manifests spasticity for at least 6 months
* Spasticity due to MS as shown by a TNmAS score equal or greater than six (≥6) in the most affected limb.
* EDSS equal or greater than 3.0
* If receiving disease-modifying medications, these must have been at a stable dose for at least three (3) months prior to screening, and the subject must be willing to maintain this treatment for the duration of the study
* Stable regimen for at least thirty (30) days prior to study entry for all medications and non-pharmacological therapies that are intended to alleviate spasticity
* Absence of infections, peripheral vascular disease, painful contractures, advanced arthritis, or other conditions that hinder evaluation of joint movement
* Have a creatinine clearance, as calculated by Glomerular Filtration Rate using the Modification of Diet in Renal Disease (MDRD) Study equation, greater than 60mL/min.
* Use of a medically highly effective of birth control during the study and for ninety (90) days thereafter for women of child-bearing potential (including female subjects and female partners of non-sterile male subjects)
* Willing to allow his or her general practitioner and consultant, if appropriate, to be notified of participation in the study

Exclusion Criteria:

* Any concomitant disease or disorder that has symptoms of spasticity or that may influence the subject's level of spasticity
* Inability to rate their level of spasticity or distinguish it from other MS symptoms
* Acute MS exacerbation requiring treatment within twelve (12) weeks of screening
* Use of intravenous methylprednisolone within the twelve (12) weeks before visit 1
* Concomitant use of medications that would potentially interfere with the actions of the study medication or outcome variables
* Use of botulinum toxin A or B within six (6) months of visit 1
* History of allergy to baclofen or any inactive component of test or reference formulation
* Pregnancy, lactation or planned pregnancy during the course of the study and for three (3) months thereafter.
* History of unstable psychiatric disease, or current signs and symptoms of significant medical disorders such as severe, progressive, or uncontrolled pulmonary, cardiac, gastrointestinal, hepatic, renal, genitourinary, hematological, endocrine, immunologic, or neurological disease
* History of seizures
* Current significant cognitive deficit, severe or untreated anxiety, severe or untreated depression
* Subjects with abnormal micturition that requires indwelling or intermittent catheterization or with lower urinary tract symptoms (LUTS) that result in a score greater than twenty-six (>26) in the Baseline USP© questionnaire
* Current malignancy or history of malignancy that has not been in remission for more than five (5) years, except effectively treated basal cell skin carcinoma
* Any other significant disease, disorder or significant laboratory finding which, in the opinion of the investigator, put the subject at risk because of participation, influence the result of the study, or affect the subject's ability to participate
* Planned elective surgery or other procedures requiring general anesthesia during the study
* Subject who is inappropriate for placebo medication in the judgment of the Investigator
* History of substance abuse within the past twelve (12) months
* Current chronic use of long acting opioids or round the clock use of short acting opioids for the treatment of pain
* Participation in another research study within thirty (30) days of Screening
* Patients who are uncooperative or unwilling to sign consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Efficacy as determined by Total Numeric Transformed Modified Ashworth scale (TNmAS) in the most affected limb. | Change in baseline from Visit 1 through Visit 9 (120 days) or end of treatment
  Change from baseline through end of treatment in the pre-dose, morning TNmAS of the most affected limb. The most affected limb is determined at baseline using the sum of scores for three major motor groups. High scores indicate more severe spasticity.
Clinical Global Impression of Change (CGIC) through end of treatment | Visit 9 (120 days) or end of study
  The CGIC is a global rating scale that captures the investigator's assessment of the subject's change in overall functional performance since starting the study. Scores range from -3 (significant worsening) to +3 (significant improvement.

SECONDARY OUTCOMES:
Changes in the Multiple Sclerosis Spasticity Scale (MSSS-88) | Baseline through Visit 9 (120 days)
  This MSSS-88 is a self-administered questionnaire for the subject to assess overall functional performance and sense of impairment with respect to the level of spasticity.
Changes in the TNmAS for the most affected limb | From baseline to visits 4 (22 days), 5 (36 days), 6 (50 days), 7 (71 days), and 9 (120 days)
  The modified Ashworth Scale is a six (6)-point rating scale that measures abnormality in tone or the resistance to passive movements. Measurements are made in three muscle groups of each limb. The most affect limb is determined at baseline, based on the sum of scores from each limb. Higher scores indicate more severe spasticity.
Changes in the TNmAS for the sum of all limbs | Baseline to visits 4 (22 days), 5 (36 days), 6 (50 days), 7 (71 days), and 9 (120 days)
  The sums of scores from all limbs are compared to the baseline sum. Higher scores indicate more severe spasticity.
Changes in Expanded Disability Status Score (EDSS) | Baseline to Visit 9 (120 Days)
  The EDSS is based on an examination by a neurologist with a scale that ranges from zero (0) to ten (10) in half point (0.5) unit increments. Higher scores represent higher levels of disability.
Changes in the Lower Extremity Manual Muscle Testing (LEMMT) Scale | Baseline to Visit 4 (22 days), Visit 5 (36 days) Visit 6 (50 days) Visit 7 (71 days) and Visit 9 (120 days)
  The LEMMT Scale is an evaluation of the function and strength of individual muscles and muscle groups based on effective performance of limb movement in relation to the forces of gravity and manual resistance. Maximum muscular strength is the maximum amount of tension or force that a muscle or muscle group can voluntarily exert in one maximal effort. Scores for each muscle or muscle group range from 0 (no detectable activity) to 5 (normal activity).
Changes in Epworth Sleepiness Scale (ESS) | Baseline to Visit 4 (22 days), Visit 5 (36 days) Visit 6 (50 days) Visit 7 (71 days) and Visit 9 (120 days)
  The ESS is used to determine the level of daytime sleepiness. The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 in eight different situations.
Changes in the subject-recorded mean daily Drowsiness Numerical Rating Scale (DNRS)score for the day prior to each visit | Baseline to Visit 4 (22 days), Visit 5 (36 days) Visit 6 (50 days) Visit 7 (71 days) and Visit 9 (120 days)
  Drowsiness will be reported by the subject using a numerical rating scale with a range of zero (0; no drowsiness) to ten (10; worst possible drowsiness). Scores will be recorded every 3 hours during the day before each designated visit.
Changes in the Urinary Symptom Profile (USP) Scale | Baseline to Visit 4 (22 days), Visit 5 (36 days) Visit 6 (50 days) Visit 7 (71 days) and Visit 9 (120 days)
  The USP is a Health-Related Quality of Life questionnaire composed of 13 items assessing urinary symptoms in adults with stress, urge, overactive bladder, or urinary obstructive symptoms.
Clinical Global Impression of Change (CGIC) | Baseline to Visit 4 (22 days), Visit 5 (36 days) Visit 6 (50 days) Visit 7 (71 days)
  The CGIC scores will be recorded at the designated intervals prior to Visit 9 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Tyle, PhD, Study Chair — Osmotica Pharmaceutical
Locations (48):
- United States (25):
  - Osmotica Study Site-138, Cullman, Alabama
  - Osmotica Site-143, Long Beach, California
  - Osmotica Study Site-123, Aurora, Colorado
  - Osmotica Study Site-110, Bradenton, Florida
  - Osmotica Study Site-142, Maitland, Florida
  - Osmotica Study Site-119, Ormond Beach, Florida
  - Osmotica Study Site-120, Pompano Beach, Florida
  - Osmotica Study Site-109, Tampa, Florida
  - Osmotica Study Site-126, Northbrook, Illinois
  - Osmotica Study Site-108, Fort Wayne, Indiana
  - Osmotica Study Site-116, Lenexa, Kansas
  - Osmotica Study Site-124, Baltimore, Maryland
  - Osmotica Study Site-136, Springfield, Massachusetts
  - Osmotica Study Site-101, Ann Arbor, Michigan
  - Osmotica Study Site-115, Johnson City, New York
  - Osmotica Study Site-113, New York, New York
  - Osmotica Study Site-141, New York, New York
  - Osmotica Study Site-125, New York, New York
  - Osmotica Study Site-106, Charlotte, North Carolina
  - Osmotica Study Site-131, Cincinnati, Ohio
  - Osmotica Study Site-127, Pittsburgh, Pennsylvania
  - Osmotica Study Site-112, San Antonio, Texas
  - Osmotica Study Site-133, Salt Lake City, Utah
  - Osmotica Study Site-129, Seattle, Washington
  - Osmotica SIte-144, Tacoma, Washington
- Russia (11):
  - Osmotica Study Site-509, Pyatigorsk, Stavropol Kray
  - Osmotica Study Site-510, Tonnel’nyy, Stavropol Kray
  - Osmotica Site-511, Krasnoyarsk
  - Osmotica Study Site-508, Krasnoyarsk
  - Osmotica Study Site-510, Krasnoyarsk
  - Osmotica Study Site-501, Moscow
  - Osmotica Study Site-502, Moscow
  - Osmotica Study Site-503, Saint Petersburg
  - Osmotica Study Site-505, Saint Petersburg
  - Osmotica Study Site-507, Saint Petersburg
  - Osmotica Study Site-506, Sestroretsk
- Ukraine (12):
  - Osmotica Study Site 614, Chernihiv
  - Osmotica Study Site-602, Dnipropetrovsk
  - Osmotica Study Site-603, Dnipropetrovsk
  - Osmotica Study Site-609, Dnipropetrovsk
  - Osmotica Study Site-611, Donetsk
  - Osmotica Study Site-613, Ivano-Frankivsk
  - Osmotica Site-605, Kharkiv
  - Osmotica Study Site-610, Kharkiv
  - Osmotica Study Site-604, Kharkiv
  - Osmotica Study Site-606, Lviv
  - Osmotica Study Site-608, Odesa
  - Osmotica Study Site-615, Uzhhorod